CLINICAL TRIAL: NCT03068026
Title: Influence of the VitaBreath Device on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Influence of the VitaBreath on Exercise Tolerance in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Tyneside General Hospital (Other Government)
Collaborators: Northumbria University (Other)
Responsible Party: Principal Investigator, Ioannis Vogiatzis, Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRC-GRA-17030-VBREATH-SH
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Non-invasive ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover trial. The two exercise modalities will be separately assessed in different groups of patients, but within each group the intervention (VitaBreath) will be compared to control (pursed-lip breathing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous exercise (Experimental): Patients will undergo a constant load exercise protocol with gas exchange analysis on a cycle ergometer. The exercise protocol will be consisted of repeated 6-min exercise bouts, separated by 2-min rest periods in between work bouts in order to allow application of the VitaBreath device. During the 1st min of each resting period participants will breathe either via the VitaBreath device or normally adopting the pursed lip breathing technique. During the 2nd min of each resting period participants will breathe normally and perform an IC maneuver to assess the magnitude of dynamic hyperinflation.
  Interventions: Device: VitaBreath; Other: Pursed Lip Breathing technique
- Interval exercise (Experimental): Patients will undergo an interval exercise protocol with gas exchange analysis on a cycle ergometer. The exercise protocol will consist of repeated 2-min exercise bouts, separated by 2-min resting periods in between work bouts in order to allow application of the VitaBreath device. During the 1st min of each resting period participants will breathe either via the VitaBreath device or normally adopting the pursed lip breathing technique. During the 2nd min of each rest period participants will breathe normally and perform an IC maneuver, to assess the magnitude of dynamic hyperinflation.
  Interventions: Device: VitaBreath; Other: Pursed Lip Breathing technique

INTERVENTIONS:
Device: VitaBreath — The VitaBreath devise will be applied during the 1st minute of each resting period between exercise bouts and during the 1st minute of recovery.
Other: Pursed Lip Breathing technique — Pursed Lip Breathing technique will be applied during the 1st minute of each resting period between exercise bouts and during the 1st minute of recovery.

SUMMARY:
People with COPD have more air in their lungs than other people (this problem with high lung volumes is called "hyperinflation"). Unfortunately this is unhelpful as breathing at higher lung volumes requires more effort and contributes to breathlessness. When anyone exercises, they breathe more quickly. People with COPD have narrowed airways, which makes breathing out difficult. When they breathe more quickly they may not be able to breathe out fully before they need to take the next breath in. This means that the volume of air in their lungs tends to increase further during exercise, which makes breathing even more difficult. This problem is called "dynamic hyperinflation".

Pulmonary rehabilitation is one of the most helpful interventions for people with COPD and most of the benefit gained is from exercise. Anything that helps people increase the amount of exercise they can perform should lead to further improvements.

Non-invasive positive pressure ventilation is a method of supporting a person's normal breathing. The ventilator delivers a flow of air at low pressure as you breathe out, which helps patients to breathe out more completely. The device also detects when patients start to breathe in and delivers a stronger flow of air at a higher pressure, helping them to take a deeper breath in. Previous research studies have shown that when people with COPD use non-invasive ventilation during exercise they are able to exercise for longer and are less breathless. The purpose of this study is to assess whether a new portable non-invasive ventilation device, called the VitaBreath, helps people with COPD recover from breathlessness during the exercise breaks more quickly (by reducing "dynamic hyperinflation", described above) and to exercise for longer overall. The VitaBreath device is small and light, weighing 0.5 kilograms (just over one pound). It is handheld and battery powered.

DETAILED DESCRIPTION:
In patients with chronic obstructive pulmonary disease (COPD) dynamic hyperinflation (DH) and the concurrent mechanical constraints on tidal volume expansion during exercise increase work of breathing and perceived respiratory discomfort, limiting endurance. An additional consequence of DH and the concomitant high mean intrathoracic pressure swings, cardiac performance and, hence, supply of oxygenated blood to the malfunctioning peripheral muscles is further compromised. This contributes to perceived leg discomfort and exercise intolerance.

Bronchodilator therapy is associated with a reduction in operating lung volumes, leading to improvements in perceived breathlessness and exercise tolerance. Heliox (helium and oxygen) is less dense and generates less airway resistance than air. Heliox breathing has been shown to improve exercise tolerance in COPD. A recent study demonstrated that compared to room air, breathing heliox during constant-load exercise (CLE) (continuous) increased inspiratory capacity (IC), and lessened DH, breathlessness and leg discomfort at isotime and at the point of exercise limitation. In addition, heliox breathing increased stroke volume, cardiac output and hence locomotor muscle oxygen delivery. However, the main drawback of heliox supplementation is the high cost, especially when it is used for long periods of time. Previous studies using inspiratory pressure support have shown improvements in dyspnoea and exercise capacity by reducing the work of breathing, as well as improved central hemodynamic responses and peripheral muscle oxygenation.

In comparison to traditional noninvasive ventilators, the Vitabreath device, which provides positive inspiratory pressure, is compact, light and inexpensive. Ease of operation, portability and battery life support use to aid relief of breathlessness, including away from the patient's home. This should facilitate maintenance of, and improvement in, activity. Vitabreath may also prove to be a useful tool to increasing exercise tolerance and the intensity of training, and hence the magnitude of physiological adaptations by mitigating DH during rehabilitative exercise training.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 40 years or older.
2. Current or previous smoking history: 10 or more pack years.
3. Spirometry confirmed stable COPD (GOLD stages II-IV) under optimal medical therapy.
4. Exhibit substantial exercise-induced dynamic hyperinflation (ΔIC baseline > 0.15 L)

Exclusion Criteria:

1. Orthopaedic, neurological or other concomitant diseases that significantly impair normal biomechanical movement patterns, as judged by the investigator.
2. Moderate or severe COPD exacerbation within 6 weeks.
3. Unstable cardiac arrhythmia.
4. Unstable ischaemic heart disease, including myocardial infarction within 6 weeks.
5. Moderate or severe aortic stenosis or hypertrophic obstructive cardiomyopathy.
6. Uncontrolled hypertension.
7. Uncontrolled hypotension (SBP<85mmHg).
8. Uncontrolled diabetes.
9. Intolerance of the VitaBreath device.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance (total exercise time) | 12 months
  The primary outcome is exercise tolerance (total exercise time) during continuous and interval exercise.

SECONDARY OUTCOMES:
Symptoms | 12 months
  Breathlessness (assessed by Borg 1-10 scale)
Dynamic hyperinflation | 12 months
  Inspiratory capacity (Litres)

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vogiatzis, Ph.D., Principal Investigator — Northumbria University of Newcastle
Locations (1):
- North Tyneside General Hospital, Newcastle upon Tyne, Northumberland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogiatzis I, Zakynthinos S. Factors limiting exercise tolerance in chronic lung diseases. Compr Physiol. 2012 Jul;2(3):1779-817. doi: 10.1002/cphy.c110015. PMID 23723024
- [Background] O'Donnell DE, Lam M, Webb KA. Spirometric correlates of improvement in exercise performance after anticholinergic therapy in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Aug;160(2):542-9. doi: 10.1164/ajrccm.160.2.9901038. PMID 10430726
- [Background] Louvaris Z, Vogiatzis I, Aliverti A, Habazettl H, Wagner H, Wagner P, Zakynthinos S. Blood flow does not redistribute from respiratory to leg muscles during exercise breathing heliox or oxygen in COPD. J Appl Physiol (1985). 2014 Aug 1;117(3):267-76. doi: 10.1152/japplphysiol.00490.2014. Epub 2014 Jun 5. PMID 24903919
- [Background] O'Donnell DE, Sanii R, Younes M. Improvement in exercise endurance in patients with chronic airflow limitation using continuous positive airway pressure. Am Rev Respir Dis. 1988 Dec;138(6):1510-4. doi: 10.1164/ajrccm/138.6.1510. PMID 3059897
- [Background] Keilty SE, Ponte J, Fleming TA, Moxham J. Effect of inspiratory pressure support on exercise tolerance and breathlessness in patients with severe stable chronic obstructive pulmonary disease. Thorax. 1994 Oct;49(10):990-4. doi: 10.1136/thx.49.10.990. PMID 7974316
- [Background] Bianchi L, Foglio K, Pagani M, Vitacca M, Rossi A, Ambrosino N. Effects of proportional assist ventilation on exercise tolerance in COPD patients with chronic hypercapnia. Eur Respir J. 1998 Feb;11(2):422-7. doi: 10.1183/09031936.98.11020422. PMID 9551748
- [Background] Wysocki M, Meshaka P, Richard JC, Similowski T. Proportional-assist ventilation compared with pressure-support ventilation during exercise in volunteers with external thoracic restriction. Crit Care Med. 2004 Feb;32(2):409-14. doi: 10.1097/01.CCM.0000108869.12426.51. PMID 14758156
- [Background] van 't Hul A, Gosselink R, Hollander P, Postmus P, Kwakkel G. Acute effects of inspiratory pressure support during exercise in patients with COPD. Eur Respir J. 2004 Jan;23(1):34-40. doi: 10.1183/09031936.03.00016903. PMID 14738228
- [Background] Rodrigues MK, Oliveira MF, Soares A, Treptow E, Neder JA. Additive effects of non-invasive ventilation to hyperoxia on cerebral oxygenation in COPD patients with exercise-related O2 desaturation. Clin Physiol Funct Imaging. 2013 Jul;33(4):274-81. doi: 10.1111/cpf.12024. Epub 2013 Jan 21. PMID 23692616
- [Background] Ambrosino N, Cigni P. Non invasive ventilation as an additional tool for exercise training. Multidiscip Respir Med. 2015 Apr 9;10(1):14. doi: 10.1186/s40248-015-0008-1. eCollection 2015. PMID 25874110